CLINICAL TRIAL: NCT05577494
Title: A Cluster Randomized Controlled Trial of Enhanced Versus Standard Measurement-Based Care Implementation for Depression
Brief Title: A Trial of Enhanced Versus Standard Measurement-Based Care Implementation for Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Children's Hospital of Fudan University (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHDC120120126
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder; Mobile Health
Keywords: major depressive disorder; measurement-based care; mobile health
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Clinicians: Three hospitals in Shanghai are included: Shanghai Mental Health Center, the Children's Hospital of Fudan University, and Tongji Hospital of Tongji university, and 100 clinicians are recruited in total. Then, they will receive an online questionnaire and complete the Clinician Questionnaire. Finally, the survey results need to be qualitatively analyzed.
  Interventions: Other: Questionnaire online
- Clinician interviewers: Three hospitals in Shanghai are included: Shanghai Mental Health Center, the Children's Hospital of Fudan University, and Tongji Hospital of Tongji university, and 30 clinicians are recruited in total (10 in each clinical institution). Each clinical institution shall select 2-3 interviewers, who shall participate in interview consistency training. Semi-structured interviews are conducted with the enrolled clinicians using the Clinician Interview Guide. The interview process needs to be recorded, and the interview results need to be qualitatively analyzed.
- Outpatients with MDD:: Three hospitals in Shanghai are included: Shanghai Mental Health Center, the Children's Hospital of Fudan University, and Tongji Hospital of Tongji university, and 600 patients with MDD are recruited in outpatient clinics (200 in each institution). The patient questionnaire will be completed online. The enrolled patients need to conduct an online questionnaire survey and complete the Patient Questionnaire. Finally, the survey results need to be qualitatively analyzed.
  Interventions: Other: Questionnaire online
- Patients with MDD receiving focus group discussion: Each center will hold 1-2 focus group symposiums for 8-10 patients according to the Patient Focus Group Symposium Manual. The content of the symposium needs to be recorded and written. Finally, the interview results need to be qualitatively analyzed.

INTERVENTIONS:
Other: Questionnaire online — Questionnaire online: all subjects will receive an online questionnaire and complete the Clinician Questionnaire.
  Semi-structured interviews: semi-structured interviews are conducted with the clinician interviewers using the Clinician Interview Guide.
  Focus group discussion: Focus group discussions are conducted with patients according to the Patient Focus Group Symposium Manual.
  Other Names: Semi-structured interviews; Focus group discussion
  Groups: Clinicians; Outpatients with MDD:

SUMMARY:
Measurement-based care (MBC) is an evidence-based practice that incorporates routine outcome assessment using validated rating scales to guide collaborative clinical decision-making. Although MBC results in improved outcomes for patients with major depressive disorder (MDD), there are barriers to its broad implementation in clinical settings. The use of "enhanced" MBC (eMBC), with mobile apps that allow patients to track outcomes and engage in self-management via WeChat, may address some of these barriers. This study intends to compare differences of efficacy between the implementation with eMBC using WeChat and the standard MBC implementation using paper-pencil assessments at the clinic, for both implementation and clinical outcomes.

DETAILED DESCRIPTION:
Measurement-based care (MBC) is an evidence-based practice that incorporates routine outcome assessment using validated rating scales to guide collaborative clinical decision-making. Although MBC results in improved outcomes for patients with major depressive disorder (MDD), there are barriers to its broad implementation in clinical settings. The use of "enhanced" MBC (eMBC), with mobile apps that allow patients to track outcomes and engage in self-management via WeChat, may address some of these barriers. Therefore, we present a trial protocol for a 2-arm cluster randomized controlled trial (RCT) with a hybrid implementation-effectiveness design comparing standard MBC implementation versus eMBC implementation with 6-month follow up in 12 mental health centers in Shanghai, China. The eMBC implementation uses a WeChat mini-program that includes outcome tracking using brief questionnaires and self-management lessons supplemented with support by a lay coach via WeChat. The primary implementation outcome is implementation reach, defined as the proportion of eligible patients with a PHQ-9 score recorded in the hospital chart at 6 months after MBC implementation. The primary clinical outcome is clinical remission, defined as a PHQ-9 score of 4 or less at the 6-month follow up. Other implementation and clinical outcomes will be examined, including medication adherence, doctor-patient alliance, and a piggy-back cost-benefit economic analysis. Qualitative interviews will be conducted with physicians and patients to produce an interpretive account of the contextual factors which impact eMBC implementation. This study intends to compare differences of efficacy between the implementation with eMBC using WeChat and the standard MBC implementation using paper-pencil assessments at the clinic, for both implementation and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for clinicians:

* Recruited clinicians who are on the job and they come from Shanghai Mental Health Center, the Children's Hospital of Fudan University, and Shanghai Tongji Hospital
* Recruited clinicians are of different ages, working years and genders;
* Recruited clinicians understand the research content and sign the informed consent form

Inclusion criteria for patients with MDD:

* Recruited patients should be definitely diagnosed as "MDD" in their outpatient records, and those patients are in a stable state of illness and can cooperate in completing the questionnaire survey or accepting the focus group discussion;
* Recruited patients have junior high school education or above, as well as adequate audio-visual skills, and can fully understand the informed consent form and interview content.
* The age of the recruited patients is 12-65 years, and the number of children and adolescents aged 12-18 years is not less than one third of the total sample size of patients;
* The enrolled patients or the guardian of them can understand the research content and sign the informed consent form.

Exclusion Criteria:

Exclusion criteria for clinicians:

* Recruited clinicians are unable to conduct effective verbal conversation;
* Recruited clinicians are unable to cooperate or complete other situations of the interview.

Exclusion criteria for patients with depression:

* Recruited patients who have obvious violent attacks or tendencies;
* Recruited patients who are in the attack or unstable period of illness;
* There is a serious tendency to commit suicide;
* Recruited patients who are unable to conduct effective verbal conversation;
* Recruited patients who cannot cooperate or complete other situation of the interview.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects of clinicians come from Shanghai Mental Health Center, the Children's Hospital of Fudan University, and Tongji Hospital of Tongji University, whose age, working years, and gender are different.
  Subjects of outpatients come from Shanghai Mental Health Center, the Children's Hospital of Fudan University, and Tongji Hospital of Tongji University who have been definitely diagnosed as MDD and are in stable condition. Their age is between 12 and 65 years old, and the number of children and adolescents aged 12 to 18 years old is not less than one third of the total sample size of patients. In addition, they have junior high school education and above, as well as adequate audio-visual skills, and can fully understand the informed consent form and interview content.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
judge the key barriers and promoting factors of the follow-up experiment implementation. | 1years, anticipated
  Through the qualitative method of focus group interviews with clinicians and patients, the specific factors hindering the implementation of eMBC by doctors and patients, and the direction of follow-up specific intervention will be identified. Through the quantitative method of online survey of doctors and patients, the population to be implemented in the following second stage, the content and frequency of full course follow-up will be determined, and the specific definition of depression on the full course model will be improved.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Chen, Study Chair — Shanghai Mental Health Center; Jinhua Sun, Study Chair — The Children's Hospital of Fudan University; Qingwei Li, Study Chair — Tongji Hospital
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China